CLINICAL TRIAL: NCT00614887
Title: Hypothalamo-, Pituitary-, Adrenal Axis Dysfunction in Subarachnoid Hemorrhage
Acronym: SAHENDO
Status: Completed | Type: Observational
Sponsor: Kuopio University Hospital (Other)
Collaborators: University of Eastern Finland (Other)
Responsible Party: Bendel Stepani, MD, Kuopio University Hospital
Other Study IDs: KUH5070184; 5070184
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Last update posted 2023-10-26 (Actual); Status verified 2008-01

CONDITIONS: Subarachnoid Hemorrhage; Cerebral Aneurysm
Keywords: Subarachnoid hemorrhage; Pituitary gland; Adrenal gland
MeSH Terms: conditions — Subarachnoid Hemorrhage; Intracranial Aneurysm; Pituitary Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum and plasma samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 2: Patients scheduled for elective cerebral aneurysmal surgery
- 1: Patients with subarachnoid hemorrhage

SUMMARY:
Subarachnoid haemorrhage (SAH) may cause damage to the hypotalamo-pituitary-adrenal axis (HPA) thus disturbing the hormonal response of these structures.

The aim of our study is to characterize the function of HPA-axis acutely and over time up to three months in patients with SAH.

DETAILED DESCRIPTION:
The hypotalamo-pituitary-adrenal (HPA)-axis may be affected in SAH by temporary or permanent damage to the hypothalamus and/or pituitary gland. Also surgery or endovascular treatment of a ruptured intracranial aneurysm may affect the hormonal response of the HPA-axis. Some data suggest a high incidence of delayed endocrine abnormalities in patients with SAH but only little data exists on the acute endocrine abnormalities in this disease.

We will study the pituitary-adrenal hormone levels in patients with acute aneurysmal SAH and patients admitted for elective cranial aneurysm surgery will serve as a control population. We will use serum free cortisol calculation and total cortisol measurements as well as adrenocorticotrophic hormone (ACTH) stimulation test in assessing the responsiveness of the adrenal gland to exogenous ACTH. The hormone levels will be measured repeatedly during the first seven days after SAH and once at three months.

ELIGIBILITY:
Inclusion Criteria:

SAH-group:

* >age 18,
* Subarachnoid hemorrhage due to an cerebral aneurysm

Control group:

* Age >18
* Admitted for elective primary cerebral aneurysm surgery

Exclusion Criteria:

SAH group:

* Any corticoid treatment (also inhaled)
* Usage of etomidate before study entry or during the study period
* Exact bleeding day unknown
* Previous history of SAH or more than three days of current bleeding
* Previous aneurysm surgery or embolization
* Traumatic SAH
* Known pituitary insufficiency and moribund state of the patient
* Refusement of the patient

control group:

* Any corticoid treatment (also inhaled)
* Usage of etomidate before study entry or during the study period
* Previous history of SAH or cerebral aneurym surgery or embolization
* Admitted for elective aneurysm embolization
* Known pituitary insufficiency
* Refusement of the patienT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from acute subarachnoid hemorrhage and patients admitted for elective aneurysm surgery.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2006-03; Primary Completion 2006-11 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stepani J Bendel, MD, Principal Investigator — Department of Intensive Care, Kuopio University Hospital, FINLAND; Ari Uusaro, MD, Phd, Study Director — Department of Intensive Care, Kuopio University Hospital, FINLAND; Timo Koivisto, MD, Phd, Study Director — Department of Neurosurgery, Kuopio Universtiy Hospital, FINLAND
Locations (1):
- Department of Intensive Care, Kuopio University Hospital, Kuopio, PL 1777, Finland

REFERENCES:
- [Derived] Bendel S, Koivisto T, Ryynanen OP, Ruokonen E, Romppanen J, Kiviniemi V, Uusaro A. Insulin like growth factor-I in acute subarachnoid hemorrhage: a prospective cohort study. Crit Care. 2010;14(2):R75. doi: 10.1186/cc8988. Epub 2010 Apr 28. PMID 20426845
- [Derived] Bendel S, Koivisto T, Ruokonen E, Rinne J, Romppanen J, Vauhkonen I, Kiviniemi V, Uusaro A. Pituitary-adrenal function in patients with acute subarachnoid haemorrhage: a prospective cohort study. Crit Care. 2008;12(5):R126. doi: 10.1186/cc7084. Epub 2008 Oct 13. PMID 18851750